CLINICAL TRIAL: NCT03843554
Title: The ARMOR Trial: Commensal Oral Microbiota as a Trigger of Oral Mucositis Severity
Brief Title: Commensal Oral Microbiota in Head and Neck Cancer
Acronym: ARMOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated with 50% enrollment by the sponsor due to under enrollment into specific diverse racial, ethnic, and sex/gender categories.
  https://grants.nih.gov/policy/inclusion/women-and-minorities.htm
Sponsor: University of Pennsylvania (Other)
Collaborators: NYU Langone Health (Other); The Forsyth Institute (Other); Medical University of South Carolina (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Patricia Corby, DDS, Associate Dean of Translational Research, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 832750; U01DE027637 (NIH); UPCC 06319 (Other: University of Pennsylvania Cancer Center)
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Oral Mucositis
Keywords: Head Cancer; Neck Cancer; Oral Mucositis; Oral Health; Radiation; Chemoradiation
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis | interventions — Dental Prophylaxis

STUDY DESIGN:
Intervention Model Description: Prospective, single blind, two arm, randomized, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors will grade the oral mucositis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Oral Hygiene (Placebo Comparator): Standard of Care Oral Hygiene group (SOC-OH): Subjects assigned to SOC-OH will attend weekly oral care visits where they will have their teeth brushed with a soft bristled toothbrush by the interventionist. No treatment to the oral mucosa will be provided to this group as part of the intervention. Subjects will receive oral care instructions and will be asked to follow SOC oral hygiene instructions at home.
  Interventions: Other: Standard of Care Oral Hygiene
- Oral Mucosal Deterging and Dental Prophylaxis (OMDP) (Experimental): Oral Mucosal Deterging & Dental Prophylaxis (OMDP) protocol: Subjects assigned to OMDP will attend weekly intervention visits during which they will have their teeth cleaned and will receive the OMDP intervention as follows: subjects will receive a professional dental prophylaxis including periodontal surface debridement and deterging of the oral mucosal surfaces. Subjects will be asked to follow OMDP oral hygiene instructions at home.
  Interventions: Procedure: Oral mucosal deterging and dental prophylaxis

INTERVENTIONS:
Other: Standard of Care Oral Hygiene — Standard of care oral hygiene- weekly oral care visits with soft-bristled toothbrushing.
  Arms: Standard of Care Oral Hygiene
Procedure: Oral mucosal deterging and dental prophylaxis — Subjects will receive a professional dental prophylaxis including periodontal surface debridement [a light-touch, gentle form of instrumentation performed with an ultrasonic instrument to promote plaque removal, to facilitate biofilm disruption and endotoxin flushing, but yet with the preservation of the periodontal cementum] and deterging of the oral mucosal surfaces.
  Arms: Oral Mucosal Deterging and Dental Prophylaxis (OMDP)

SUMMARY:
The ARMOR Trial will test the efficacy of an oral care protocol to treat oral mucositis (OM) in patients receiving radiation (RT) or chemoradiation (chemoRT) for head and neck cancer. Participants will attend a screening/baseline visit, weekly intervention visits while they are undergoing RT or chemoRT, and a visit 3 months after completing RT or chemoRT. At intervention visits, samples will be collected (such as saliva, oral swabs) and participants will receive their assigned study intervention, either Oral Mucosal Deterging and Dental Prophylaxis protocol (OMDP), which includes a dental cleaning and treatment to the oral mucosa, or a Standard of Care Oral Hygiene, which includes teeth brushing and no treatment to the oral mucosa.

DETAILED DESCRIPTION:
This is a prospective, single blind, two arm, randomized, controlled trial to test the efficacy of an oral care protocol to treat oral mucositis (OM) in patients receiving radiation (RT) or chemoradiation (chemoRT) for head and neck cancer. This trial will also measure salivary proinflammatory cytokines, and evaluate other clinical effects of the intervention during cancer therapy. In addition, oral mucosal swabs will be collected for the future characterization of changes in the microbiome associated with OM severity.

Patients will be randomized in a 1:1 ratio to two different oral care protocols within 4 strata defined by type of RT (Proton beam therapy (Protons)) vs intensity-modulated radiation therapy (IMRT) and cancer treatment (RT versus chemoRT). Eligible subjects will be assigned to receive either the Oral Mucosal Deterging and Dental Prophylaxis protocol (OMDP) or a Standard of Care Oral Hygiene protocol (SOC-OH). Prior to randomization, all enrolled subjects will receive a baseline dental prophylaxis and fluoride varnish application prior to start of RT or chemoRT to ensure that all subjects enter the study with comparable oral health. Subjects assigned to OMDP will receive the OMDP Protocol (Oral Mucosal Deterging and Dental Prophylaxis) at weekly intervention visits. Subjects randomized to the SOC-OH will receive oral health instructions following the American Dental Association Guidelines and will have their teeth cleaned (brushed) during weekly intervention visits; no treatment to the oral mucosa will be provided to this group.

At each bi-weekly study visit, study assessments will include the collection of saliva and oral mucosal swabs, an oral exam and OM assessment, and the completion of questionnaires. During the course of the study, subjects will attend one baseline visit, up to 9 intervention visits, and a follow-up visit approximately 3 months after completion of RT. Local supportive care, including normal saline rinses, topical anesthetics, mixed medication mouthwashes (e.g. Magic Mouthwash), feeding tubes, and pain management will be allowed according to each recruitment site's standard of care procedures.

ELIGIBILITY:
Currently enrolling subjects receiving intensity-modulated radiation therapy (IMRT), with or without chemotherapy.

Subject Inclusion Criteria

To participate in this study, an individual must meet all the following criteria:

1. 18 years of age or older;
2. Able and willing to provide informed consent prior to initiation of study procedures;
3. Scheduled to undergo radiation or chemoradiation treatment for head/neck cancer;
4. Presents with at least one of nine areas of the oral or oropharyngeal mucosa (i.e., upper lip, lower lip, right cheek, left cheek, right ventral and lateral tongue, left ventral and lateral tongue, floor of the mouth, and soft palate) expected to receive at least 5000 cGy of RT. Patients with cancer located outside of the oral cavity will be included when at least 5000 cGy of RT will be administered to the oral cavity in addition to the RT targeted at the primary cancer site.
5. Presents with a minimum of 6 natural teeth.

Subject Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnant or lactating at the baseline/screening visit;
2. Participating in another oral health interventional research study at any point during their participation in this trial;
3. Receiving induction chemotherapy or concurrent radiation therapy with cetuximab;
4. Reports current use of antifungal or antibiotic at the time of enrollment;
5. Presents with immunocompromised status (defined as an absolute neutrophil count (ANC) of less than 1000);
6. Presents with any of the following conditions, which based on American Dental and American College of Cardiology guidelines, require antibiotic prophylaxis prior to dental treatment:

   1. prosthetic cardiac valves, including transcatheter-implanted prostheses and homografts;
   2. prosthetic material used for cardiac valve repair, such as annuloplasty rings and chords;
   3. a history of infective endocarditis;
   4. a cardiac transplant with valve regurgitation due to a structurally abnormal valve;
   5. the following congenital (present from birth) heart disease: unrepaired cyanotic congenital heart disease, including palliative shunts and conduits; or any repaired congenital heart defect with residual shunts or valvular regurgitation at the site of or adjacent to the site of a prosthetic patch or a prosthetic device;
7. Presents with cardiovascular implantable electronic devices (CIEDs) such as pacemakers, and implantable cardioverter-defibrillators; unless, a) in the opinion of the investigator, the OMDP protocol can be performed with hand scalers (and not with an ultrasonic device as per protocol) or upon consult with the treating cardiologist, it is determined that the ultrasonic device can be safely used;
8. Presents with severe periodontal disease for which treatment cannot be completed prior to the start of radiation/chemoradiation (at the discretion of the investigator);
9. Had surgery as part of cancer treatment and is not sufficiently healed to comply with study requirements prior to RT initiation;
10. In the opinion of the investigator, is unable or unlikely to comply fully with the study requirements or procedures for any reason (e.g. cognitive or physical impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Corby, DDS, Principal Investigator — University of Pennsylvania; Alex Lin, MD, Principal Investigator — Penn Medicine, Perelman Center for Advanced Medicine
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: H&N cancer patients were recruited to achieve 120 study subjects. The primary recruitment of 60 subjects was done through the UPenn Cancer Center.
  The sponsor/NIDCR prematurely ceased enrollment in proton therapy. Afterwards, the sponsor terminated the trial with 50% enrollment due to "under-enrollment into specific diverse racial, ethnic, and sex/gender categories." As a result, the analysis are presented for all randomized subjects (30 per arm).
Groups:
- Oral Mucosal Deterging and Dental Prophylaxis (OMDP): Oral Mucosal Deterging & Dental Prophylaxis (OMDP) protocol: Subjects assigned to OMDP will attend weekly intervention visits during which they will have their teeth cleaned and will receive the OMDP intervention as follows: subjects will receive a professional dental prophylaxis including periodontal surface debridement and deterging of the oral mucosal surfaces. Subjects will be asked to follow OMDP oral hygiene instructions at home.
  Oral mucosal deterging and dental prophylaxis: Subjects will receive a professional dental prophylaxis including periodontal surface debridement [a light-touch, gentle form of instrumentation performed with an ultrasonic instrument to promote plaque removal, to facilitate biofilm disruption and endotoxin flushing, but yet with the preservation of the periodontal cementum] and deterging of the oral mucosal surfaces].
Period: Overall Study
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP)
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: ARMOR Trial employed a two-arm (OMDP vs STANDARD) parallel group design. Data were available on 30 subjects in each arm who received IMRT treatment (n=60). Baseline characteristics and demographics were presented for all 60 randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants] — Population: The ARMOR Trial employed a two-arm (OMDP vs STANDARD) parallel group design. The goal was to randomize 120 subjects within the 4 strata defined by planned cancer treatment (IMRT versus Proton, with or w/o chemotherapy). The first subject was randomized on 10/11/2019. On 2/19/2021, the study team received a NIDCR/DSMB letter recommending discontinuing enrollment for subjects receiving Proton beam therapy. The trial was closed by the NIDCR on 08/03/22.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 19 | 25 | 44
    >=65 years | 11 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The ARMOR Trial employed a two-arm (OMDP vs STANDARD) parallel group design. The goal was to randomize 120 subjects within the 4 strata defined by planned cancer treatment (IMRT versus Proton, with or w/o chemotherapy). The first subject was randomized on 10/11/2019. On 2/19/2021, the study team received a NIDCR/DSMB letter recommending discontinuing enrollment for subjects receiving Proton beam therapy. The trial was closed by the NIDCR on 08/03/22.
  years | 61.9 (7.6) | 58.1 (8.4) | 60.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The ARMOR Trial employed a two-arm (OMDP vs STANDARD) parallel group design. The goal was to randomize 120 subjects within the 4 strata defined by planned cancer treatment (IMRT versus Proton, with or w/o chemotherapy). The first subject was randomized on 10/11/2019. On 2/19/2021, the study team received a NIDCR/DSMB letter recommending discontinuing enrollment for subjects receiving Proton beam therapy. The trial was closed by the NIDCR on 08/03/22.
  Participants
    Female | 4 | 2 | 6
    Male | 26 | 28 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ARMOR Trial employed a two-arm (OMDP vs STANDARD) parallel group design. The goal was to randomize 120 subjects within the 4 strata defined by planned cancer treatment (IMRT versus Proton, with or w/o chemotherapy). The first subject was randomized on 10/11/2019. On 2/19/2021, the study team received a NIDCR/DSMB letter recommending discontinuing enrollment for subjects receiving Proton beam therapy. The trial was closed by the NIDCR on 08/03/22.
  Participants
    Hispanic or Latino | 2 | 1 | 3
    Not Hispanic or Latino | 28 | 29 | 57
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ARMOR Trial employed a two-arm (OMDP vs STANDARD) parallel group design. The goal was to randomize 120 subjects within the 4 strata defined by planned cancer treatment (IMRT versus Proton, with or w/o chemotherapy). The first subject was randomized on 10/11/2019. On 2/19/2021, the study team received a NIDCR/DSMB letter recommending discontinuing enrollment for subjects receiving Proton beam therapy. The trial was closed by the NIDCR on 08/03/22.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 29 | 27 | 56
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Oral Mucosal Severity (Grade 3 or 4)
Description: World Health Organization's Oral Toxicity Scale (WHO OTS): Oral mucositis severity as measured by the WHO OTS; severity is graded 0 through 4, with 4 being the worst. Grade 0 (none), Grade 1 (oral soreness, erythema), Grade 2 (ulceration, solid diet tolerated), Grade 3 (ulceration, liquid diet only), and Grade 4 (nothing by mouth).
Time Frame: Week 1 (Day 0/Randomization) - Week 8 (Day 56) during radiation therapy. Change from Baseline to Final Intervention Visit (FIV) is the endpoint being analyzed at this single timepoint (Day 56 relative to Day 0).
Population: 60 randomized subjects, 30 per arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP)
Number analyzed (Participants) | 30 | 30
Participants | 9 | 8
Statistical Analysis 1: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); Test type: Superiority — Primary hypothesis. Null hypothesis is that the proportion of patients with a successful outcome of WHO OM severity grades 0-2 at the post study evaluation will not differ between the two randomized intervention groups. The estimated proportion of successes from our pilot trial is 0.30 with SOC. The alternative hypothesis is that the proportion of patients with a successful outcome differs between the two groups from the SOC proportion of 0.30 by +/-0.265 or more; p = 0.999, Fisher Exact; OM WHO grading scale (less or equal to 2) severity employed a two-sided Fisher's exact test to compare the two arms at Visit 9

2. Secondary Outcome: Inflammatory Markers Correlative Measures
Description: Salivary cytokines: Levels of Th1/Th2-type cytokines IL10, IL8, IL12p70, TNF alpha, IL4, IL1b, IL2, IL13, IL5, and IFN gamma will be assessed, in addition to levels of gp340.
Time Frame: Baseline and final intervention visit.
Population: Inflammation markers were summarized by treatment group, visit and sample type using standard descriptive statistics. The impact of each treatment arm on the change from Baseline to Final Intervention Visit (FIV) for the above inflammation markers was examined and inferential tests such as two-sided t-test (for continuous inflammation scores change).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP)
Number analyzed (Participants) | 30 | 30
pg/mL
  IL1a | 53.9 (84.4) | 50.6 (152.9)
  IL1b | 30.4 (26.5) | 13.3 (44.9)
  IL2 | 37.9 (39.2) | -64.3 (249.8)
  IL4 | 7.7 (30.0) | -12.7 (34.9)
  IL5 | 2.2 (6.5) | 0.5 (8.5)
Statistical Analysis 1: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); The change in the inflammatory marker from baseline to the final intervention visit was analyzed using 95% confidence intervals and presented by treatment group. The two-sided t-test was used to compare the change in inflammatory markers between the two groups; Test type: Superiority — OMDP-STANDARD; p = 0.6336, t-test, 2 sided — The above t-test p-value is for IL1a; Mean Difference (Final Values) = -3.3, Standard Error of Mean 174.6
Statistical Analysis 2: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); The change in the inflammatory marker from baseline to the final intervention visit was analyzed using 95% confidence intervals and presented by treatment group. The two-sided t- test was used to compare the change in inflammatory markers between the two groups; Test type: Superiority — OMDP-STANDARD; p = 0.3510, t-test, 2 sided — IL1b; Mean Difference (Final Values) = -17.1, Standard Error of Mean 52.1
Statistical Analysis 3: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); [analysis description as in outcome 2, analysis 2]; Test type: Superiority — OMDP-STANDARD; p = 0.3510, t-test, 2 sided — IL2; Mean Difference (Final Values) = -102.2, Standard Error of Mean 252.8
Statistical Analysis 4: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); [analysis description as in outcome 2, analysis 2]; Test type: Superiority — IL4; p = 0.8371, t-test, 2 sided; Mean Difference (Final Values) = -20.4, Standard Error of Mean 46.0
Statistical Analysis 5: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); [analysis description as in outcome 2, analysis 2]; Test type: Superiority — IL5; p = 0.2991, t-test, 2 sided; Mean Difference (Final Values) = -1.7, Standard Error of Mean 10.7

3. Secondary Outcome: Duration of OM Severity
Description: OM severity (Grade 3 or more) was measured by a blinded member of the study team using the WHO OTS (previously described) and the duration and time to onset of severe OM measured in days.
Time Frame: Baseline and visits 1-9 interval during radiation therapy (area under the curve).
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP)
Number analyzed (Participants) | 30 | 30
weeks | 0.667 [0.125 to 2.056] | 0.433 [0.052 to 1.61]
Statistical Analysis 1: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); Test type: Superiority — OMDP-STANDARD; p = 0.2373, t-test, 2 sided; Mean Difference (Final Values) = -0.2293, 95% CI 2-sided [-1.9060 to 1.4475], Standard Error of Mean 0.8555

4. Secondary Outcome: Salivary Hypofunction
Description: Saliva flow rate (mL/minute) from baseline to subsequent visits was assessed by a 5-minute stimulated saliva collection. The outcome analyzed was the change from baseline to subsequent visits in saliva.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/minute
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP)
Number analyzed (Participants) | 30 | 30
mL/minute | -0.878 (0.0822) | -0.821 (0.0822)
Statistical Analysis 1: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); Test type: Superiority — OMDP-STANDARD; p = 0.6263, ANCOVA — A Week 8 general linear mixed effects model (GLM) was used to compare the change in saliva flow rate from Baseline (day 0) to week 8 (day 56) between the two groups. The change was calculated by subtracting week 8 saliva flow rate from the Baseline; Mean Difference (Final Values) = 0.0569, 95% CI 2-sided [-0.1755 to 0.2893], Standard Error of Mean 0.1160 — Estimation of the difference in least-square means for the change from Baseline to FIV in saliva flow rate

5. Secondary Outcome: Pain Scores
Description: The average pain of OM was measured subjectively (visual analog scale 0-10) and obtained by having subjects complete a questionnaire with questions based on an eleven-point numeric scale regarding oral pain (0 being no pain and 10 being maximum pain).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: 0-10 score on a scale
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP)
Number analyzed (Participants) | 30 | 30
0-10 score on a scale | -7.39 (3.51) | 5.45 (3.43)
Statistical Analysis 1: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); Test type: Superiority — OMDP-STANDARD; p = 0.6956, Regression, Linear; A Week 8 (Day 56) GLM analyzing the pain change Week 8 relative to Baseline (Day 0) was used with treatment and Baseline pain as covariates; Mean Difference (Net) = -1.94 — Difference in least-square mean change from baseline to Visit 9 in pain score

6. Secondary Outcome: QOL and Function
Description: Quality of life and function was assessed using the validated EORTC-QLQ-C30 for head and neck cancers. This questionnaire assesses general quality of life as well as issues specific to head and neck cancer patients (e.g. difficulty swallowing, pain, dry mouth). The analysis was focused on EORTC-QLC30 Questions 31 through 48. High scores indicate better QOL. High scores for the Sypmton Scale are indicative of deterioration.
Time Frame: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: 0-100 score on a scale
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP)
Number analyzed (Participants) | 30 | 30
0-100 score on a scale | 0.323 [0.1520 to 0.494] | 0.135 [-0.0333 to 0.303]
Statistical Analysis 1: Comparison: Standard of Care Oral Hygiene vs Oral Mucosal Deterging and Dental Prophylaxis (OMDP); The statistical analysis comprised an ANCOVA for a longitudinal response based on a generalized linear mixed effects repeated measures model (GLMER). The response variable is the mean change from Baseline to Visit 9 in EORTC QLQ-C30 Questions 31-48 (total); Test type: Superiority — OMDP-STANDARD; p = 0.1153, ANCOVA; ANCOVA via generalized linear mixed repeated measures model (GLMER); Mean Difference (Final Values) = -0.188, 95% CI 2-sided [-0.4095 to 0.0334], Standard Error of Mean 0.1130

ADVERSE EVENTS:
Time Frame: Percentages and numbers of participants were used to summarize AEs and SAEs. AEs record all related adverse events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation in source documents. At each study visit, the investigator inquired about the occurrence of AE/SAEs since the last visit. Events were followed for outcome information until resolution or stabilization.
Description: Serious Adverse Events: 5 subjects in Arm 1 and 0 subjects in Arm 0 experienced an AE graded as severe. 4 of those AE's were also classified as serious. No serious adverse events were determined to be related to the study treatment and/or procedures.
Groups:
- Standard of Care Oral Hygiene: Standard of Care Oral Hygiene group (SOC-OH): Subjects assigned to SOC-OH will attend weekly oral care visits where they will have their teeth brushed with a soft bristled toothbrush by the interventionist. No treatment to the oral mucosa will be provided to this group as part of the intervention. Subjects will receive oral care instructions and will be asked to follow SOC oral hygiene instructions at home. Standard of Care Oral Hygiene: Standard of care oral hygiene- weekly oral care visits with soft-bristled toothbrushing.
Arm/Group | Standard of Care Oral Hygiene | Oral Mucosal Deterging and Dental Prophylaxis (OMDP)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 5/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Oral Hygiene (N=30) | Oral Mucosal Deterging and Dental Prophylaxis (OMDP) (N=30)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Initial or prolonged hospitalization
Cholangiocarcinoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neck mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adult failure to thrive (Social circumstances) | 1 (1) | 0 (0) — Initial or prolonged hospitalization
Gout acute (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The goal was to randomize 120 subjects within the 4 strata defined by planned cancer treatment (IMRT versus Proton, with or w/o chemotherapy). The first subject was randomized on 10/11/2019. On 2/19/2021, the NIDCR/DSMB recommended to discontinue enrollment in the Proton arm. The trial was terminated on 08/31/22. Study was terminated with 50% enrollment by the sponsor due to -under enrollment into specific diverse racial, ethnic, and sex/gender categories. Only IMRT cases were used for analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT03843554/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT03843554/SAP_001.pdf